CLINICAL TRIAL: NCT05590442
Title: Early Diagnosis and Risk Evaluation of Mild Cognitive Impairment in Diabetes
Brief Title: Risk Model of Cognitive Impairment in Diabetes
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: MCImodel2022
Record Dates: First submitted 2022-09-14; First posted 2022-10-21 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes Mellitus; Mild Cognitive Impairment
Keywords: Cognitive Assessments; Olfactory Test; Risk Model
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: The patients will be divided into the training and validation cohorts with a ratio of 7:3. The training cohort will be used to screen variables and construct the model.
  Interventions: Other: Tests
- Validation cohort: The validation cohort will be used to validate the results obtained using the training cohort.
  Interventions: Other: Tests

INTERVENTIONS:
Other: Tests — Cognitive assessments and olfactory tests

SUMMARY:
Development and validation of a risk model for predicting the risk of mild cognitive impairment among individuals of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus ;
* Aged:40 -80 years ;
* Montreal Cognitive Assessment Scale (MoCA) scores 19 - 30;

Exclusion Criteria:

* Mini-mental State Examination(MMSE) scores < 24;
* Other dementia related neurological diseases or depression, schizophrenia in the past 2 years;
* Central nervous system diseases, including brain trauma, intracranial hemorrhage, acute cerebral infarction;
* Severe sinusitis, nasal cavity and sinus polyps, skull base or nasopharyngeal tumors and other space occupying lesions, congenital diseases and traumatic history of nose, maxillofacial and skull base affecting olfaction;
* Diabetic acute and chronic complications, including diabetic ketoacidosis, a hyperglycemic hyperosmolar state or severe hypoglycemic coma.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The rate of mild cognitive impairment occurrence | 1 year
  The rate of Montreal Cognitive Assessment(MoCA) scores less than 26 points after 1 year's follow-up.

SECONDARY OUTCOMES:
Glycaemic control measured by blood test. | 1 day
  HbA1c
Physical assessments. | 1 day
  BMI(body mess index) in kg/m^2
Olfactory threshold test | 1 day
  The same odor with 2 different concentrations are given to the participant each time to find out which one is more intense. (Olfactory software will analyse and give threshold score depending on participant's choice.)
Olfactory memory test | 1 day
  PART A: Participants are shown 4 pictures for each odor(10 odors in total). They select what they sniffed.
  10 minutes break. PART B: Participants sniff 20 different odors , 10 of which are same odors in PART A. They select the picture and figure out whether the odor is old or new.
Montreal Cognitive Assessment (MoCA) score | 1 day
  The MoCA is a cognitive screening test designed to assist health professionals in detection of mild cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Zhang W, Zhu D, Bi Y. Olfactory Dysfunction Mediates Adiposity in Cognitive Impairment of Type 2 Diabetes: Insights From Clinical and Functional Neuroimaging Studies. Diabetes Care. 2019 Jul;42(7):1274-1283. doi: 10.2337/dc18-2584. Epub 2019 May 21. PMID 31221697
- [Background] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Lu J, Bi Y, Zhu D. Altered Odor-Induced Brain Activity as an Early Manifestation of Cognitive Decline in Patients With Type 2 Diabetes. Diabetes. 2018 May;67(5):994-1006. doi: 10.2337/db17-1274. Epub 2018 Mar 2. PMID 29500313
- [Background] Cheng H, Zhang Z, Zhang B, Zhang W, Wang J, Ni W, Miao Y, Liu J, Bi Y. Enhancement of Impaired Olfactory Neural Activation and Cognitive Capacity by Liraglutide, but Not Dapagliflozin or Acarbose, in Patients With Type 2 Diabetes: A 16-Week Randomized Parallel Comparative Study. Diabetes Care. 2022 May 1;45(5):1201-1210. doi: 10.2337/dc21-2064. PMID 35263425